CLINICAL TRIAL: NCT07147634
Title: Outdoor Science Education and Child Well-being in Primary Schools: Protocol for a Cluster Randomized Controlled Trial on Learning, Connection to Nature, Eco-anxiety, and Stress
Acronym: Bio-Explo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Philippe Ayotte-Beaudet, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-3453; 435-2022-0651 (Other Grant/Funding Number: Social Sciences and Humanity Research Council (Canada))
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Children
Keywords: Stress; School-Based Intervention; Cluster Randomized Controlled Trial; Primary School; Connection to Nature; Eco-anxiety; Science Learning; Outdoor Education

STUDY DESIGN:
Intervention Model Description: The science education intervention consists of teaching Québec's mandatory science curriculum, focusing on life science topics and issues.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor science education (Experimental): 2h of outdoor science education intervention per week for a total of 5 weeks (following Québec's mandatory curriculum)
  Interventions: Behavioral: Outdoor science education
- Indoor classroom-based science education (Active Comparator): 2h of indoor science education intervention per week for a total of 5 weeks (following Québec's mandatory curriculum)
  Interventions: Behavioral: Indoor classroom-based science education

INTERVENTIONS:
Behavioral: Outdoor science education — Following Québec's mandatory curriculum, primary school teachers will provide life science lessons 2h/week for a total of 5 weeks in an outdoor setting
  Arms: Outdoor science education
Behavioral: Indoor classroom-based science education — Following Québec's mandatory curriculum, primary school teachers will provide life science lessons 2h/week for a total of 5 weeks inside the classroom
  Arms: Indoor classroom-based science education

SUMMARY:
The goal of this randomized controlled trial is to learn if an outdoor science education intervention can improve primary school students' learning and well-being when compared to an indoor classroom-based science education intervention. The main questions it aims to answer are:

* Will students who engage in outdoor science learning produce higher-quality observations of living organisms than students who receive instruction exclusively in an indoor, classroom-based context, when both groups are invited to make observations in an unfamiliar natural environment?
* Does an outdoor education intervention embedded within the science curriculum contribute to children's connection to nature, eco-anxiety and stress?

Participants will:

* Receive a science education intervention 2h/week for a total of 5 weeks, either indoors or outdoors
* Answer questionnaires before and after the intervention
* Participate in a field day-trip after the intervention where they will be asked to observe living organisms.

ELIGIBILITY:
Inclusion Criteria:

* Primary schools need to have a deprivation index equal to or superior to 1 (with 10 being the maximum) and be located in Montreal, Longueuil or Laval (QC).
* Teachers have to show some interest in outdoor education but are not obliged to have already done some before in order to be included.
* Only 5th and 6th grade teachers are included.
* Primary schools with two teachers interested in participating in the project.

Exclusion Criteria:

* Alternative schools or those welcoming recently arrived non-Francophone students are not included.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Score on the Scientific Observation Skills Rubric (0-15) in a Novel Environmental Context | After the 5-week intervention has ended, students will spend one day in a new environmental context (at the end of October) in order to make observations
  Students' scientific observation skills will be assessed using a structured observation rubric designed for elementary science education. After the 5-week intervention, each student will spend one day in a new environmental context (field activity at the end of October). Students will be asked to make a total of five oral observations of living organisms in this setting. Independent raters, trained in the use of the rubric, will evaluate the quality of each scientific observation using a four-level scoring framework, with scores ranging from 0 (lowest) to 3 (highest quality of scientific observation). The total score will range from 0 to 15, with higher scores indicating stronger scientific observation skills. Inter-rater agreement will be monitored to ensure reliability.

SECONDARY OUTCOMES:
Connection to nature - Score on the Inclusion of Nature in Self Scale (0-7) | At baseline and immediately after the 5-week intervention has ended
  Students' connection to nature will be assessed using the Inclusion of Nature in Self Scale (Schultz, 2001, as used in Braun & Dierkes, 2016), a validated 1-item self-report questionnaire appropriate for culturally and ethnically diverse samples of children. The item is rated on a 7-point scale (1 = nature and self do not overlap at all to 7 = nature and self completely overlap). The total score ranges from 0 to 7, with higher scores indicating a stronger subjective connection to nature. The Inclusion of Nature in Self Scale will be administered at baseline and again immediately after the 5-week intervention.
Score on the Perceived Stress Scale for Children (PSS-C; range 0-39) | At baseline and immediately after the 5-week intervention has ended
  Students' perceived stress will be assessed using the Perceived Stress Scale for Children (PSS-C), which is a standardized 13-item self-report questionnaire previously tested on a sample of Canadian children (White, 2014). Each item is rated on a 4-point Likert scale (0 = never to 3 = a lot). Scores are summed to produce a total ranging from 0 to 39, with higher scores indicating greater perceived stress. The questionnaire will be administered in class at baseline and immediately after the 5-week intervention.
Score on the 11-item Hogg Eco-Anxiety Scale (HEAS-13; range 0-33) | At baseline and immediately after the 5-week intervention has ended
  Students' eco-anxiety will be assessed using the Hogg Eco-Anxiety Scale (HEAS-13; Hogg et al., 2021), a validated 11-item self-report questionnaire. Each item is rated on a 4-point Likert scale (0 = never to 3 = almost every day). Scores are summed to produce a total ranging from 0 to 33, with higher scores indicating greater subjective feelings of eco-anxiety. The HEAS-13 will be administered in class at baseline and immediately after the 5-week intervention.
Score on the Basic Psychological Needs Satisfaction Scale - School Version (range 0-36) | Baseline and immediately after the 5-week intervention
  Students' satisfaction of the three basic psychological needs identified by Self-Determination Theory (autonomy, competence, and relatedness) will be assessed with a 9-item version of the Basic Psychological Needs Satisfaction Scale, adapted for children. Each item is rated on a 5-point Likert scale (0 = almost never to 4 = almost always). Total scores range from 0 to 36, with higher scores indicating greater satisfaction of basic psychological needs.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Ayotte-Beaudet, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Greater Montreal area (Laval, Longueuil, Montreal), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations and to protect participant confidentiality, no de-identified individual participant data will be made available. Only aggregate results will be published.